CLINICAL TRIAL: NCT07288177
Title: A Phase 2, Open-label, Multicohort Study of Rinatabart Sesutecan (Rina-S) in Participants With Non-Small Cell Lung Cancer
Brief Title: Study to Assess the Efficacy and Safety of Rina-S in Participants With Non-small Cell Lung Cancer
Acronym: RAINFOL-05
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCT1184-05; 2025-522107-18-00 (EU CTIS Number); jRCT2041250176 (Registry Identifier: Japan Registry for Clinical Trials (jRCT))
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Masking Description: Cohorts A and B will be randomized by dose. Randomization will not be used for Cohorts C, D, or E.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rina-S (Experimental): Multiple cohorts (Cohorts A, B, C, D, and E) will receive Rina-S as monotherapy.
  Interventions: Drug: Rina-S

INTERVENTIONS:
Drug: Rina-S — Intravenous (IV) infusion.
  Other Names: Rinatabart Sesutecan; PRO1184; GEN1184

SUMMARY:
This Phase 2 study will be conducted in different countries around the world with up to about 240 participants.

The purpose of this study is to evaluate how well Rina-S works against lung cancer.

The treatment in this study is Rina-S monotherapy (by itself). All participants will receive active drug; no one will be given placebo.

The treatment duration will be different for every participant, but an average of 12 months is expected. Participants will be asked to attend 1 to 5 visits at the study clinic for each cycle (duration of cycle is 3 weeks). If a participant's cancer stays the same or gets better, and there are not any serious problems, participants can keep getting study treatment for as long as the study is open.

Participation in the study will require visits to the study site(s). During site visits, there will be various tests (such as blood draws) and procedures (such as recording of heart activity, imaging/X-rays) to monitor whether the study treatment is safe and effective.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, multicenter, multi-cohort trial to evaluate the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics of Rina-S as monotherapy in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC), with or without select genomic aberrations.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has histologically or cytologically confirmed metastatic or locally advanced NSCLC of adenocarcinoma histology, not amenable to curative surgery or radiotherapy.
* Participant must have radiological disease progression while on or after receiving the most recent regimen.
* Participants either may have actionable genetic alterations (AGAs) or no AGAs.
* Participant has measurable disease according to RECIST v1.1.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1 within 7 days of Cycle 1 Day 1.

Key Exclusion Criteria (all study cohorts):

* Participant has NSCLC with histology other than adenocarcinoma
* Participant has a past or current malignancy other than the inclusion diagnosis before the planned first dose of trial treatment, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death (eg, 5-year OS ≥ 90%), including, but not limited to, adequately treated cervical carcinoma of stage 1B or less, in situ basal cell or squamous cell skin carcinoma, in situ bladder cancer, ductal carcinoma in situ, or any past malignancy considered cured for ≥ 3 years.
* Participants with newly identified or known unstable (eg, progressing brain metastases) or symptomatic central nervous system (CNS) metastases or history of carcinomatous meningitis (also known as leptomeningeal disease). Participants with history of spinal cord compression (from disease). Participants with previous CNS-directed therapy (eg, radiotherapy and/or surgery) for brain metastases may participate provided lesion(s) are radiologically stable (ie, without evidence of progression) for at least 28 days by repeat imaging.

Note: Other protocol-defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2027-11-22 (Estimated); Study Completion 2028-11-22 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as Assessed by Investigator | Approximately 3 years

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST v1.1 as Assessed by Investigator | Approximately 4 years
Disease Control Rate (DCR) per RECIST v1.1 as Assessed by Investigator | Approximately 4 years
Progression-free Survival (PFS) | Approximately 4 years
Overall Survival (OS) | Approximately 4 years
Maximum (Peak) Observed Serum Drug Concentration (Cmax) of Rina-S Related Analytes | Approximately 12 months
Time to Reach Maximum (Peak) Serum Drug Concentration (Tmax) of Rina-S Related Analytes | Approximately 12 months
Number of Participants with Antidrug Antibodies (ADAs) | Approximately 12 months
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (2):
- Virginia Cancer Specialists, Fairfax, Virginia, United States
- Japan Community Health Care Organization Chukyo Hospital, Nagoya, Minami Ward, Japan

IPD SHARING:
Plan to Share IPD: No